CLINICAL TRIAL: NCT06537752
Title: A Multi-center, Prospective, Observational stuDy to Evaluate EThanOl-induced Symptoms and Safety in Breast Cancer Patients witH Neoadjuvant/Adjuvant Chemotherapy Including Non-ethanol Formulation Docetaxel Before and After Surgery
Brief Title: A Study to Evaluate Ethanol-induced Symptoms and Safety in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-DTX-OS-402
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate ethanol-induced symptoms and safety in breast cancer patients with neoadjuvant/adjuvant chemotherapy including Non-ethanol formulation docetaxel before and after surgery

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily signed a written personal information collection and usage agreement after receiving an explanation about the objective and method, etc. of this clinical study.
* Those are confirmed to have primary breast cancers through histological diagnosis and one of the following are applicable.

  * Those who need neoadjuvant chemotherapy as breast cancer patients
  * Those who need adjuvant chemotherapy after breast cancer surgery
* Those who are scheduled to administer non-ethanol formulation docetaxel according to chemotherapy
* Those able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion.

Exclusion Criteria:

* Those are diagnosed with other primary cancer that can influence the treatment or prognosis of primary breast cancers.
* Those are diagnosed with secondary breast cancers.
* Those with Stage 0/1 (Tis, N0, M0) or Stage IV (any T, Any N, M1) breast cancers.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Breast cancer patients in need of neoadjuvant/adjuvant chemotherapy including Non-ethanol formulation docetaxel before and after surgery
Sampling Method: Non-Probability Sample
Enrollment: 1052 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of ethanol-induced symptoms in the initial cycle | From the time of treatment started until the end of follow-up(30 minutes after the treatment)
  This outcome's definition is an increase from baseline in the number of ethanol-induced symptoms during or within 30 minutes after the treatment. The initial cycle of non-ethanol formulation docetaxel is collected as 1 cycle.

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Chung-Ang University Hospital, Seoul
  - Uijeongbu Eulji Medical Center, Eulji University, Uijeongbu-si